CLINICAL TRIAL: NCT06750900
Title: Visual Feedback Manipulation in Virtual Reality Alters Movement-evoked Pain Perception in Chronic Low Back Pain
Brief Title: Visual Feedback Manipulation in Virtual Reality Alters Extension-evoked Pain Perception in Chronic LBP
Acronym: CLEVER BODY
Status: Completed | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Chair Profesor, Cardenal Herrera University
Other Study IDs: Cardenal Herrera University 67; PID2020-115609RB-C22 (Other Grant/Funding Number: MINISTRY OF SCIENCE AND INNOVATION OF SPAIN)
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Chronic Low-back Pain (cLBP)
Keywords: chronic low back pain; virtual reality; ilusions; movement-evoked pain; visual-proprioceptive feedback

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NORMAL CONDITION: The normal condition is measured as a lumbar extension without VR until the onset of pain.
  Interventions: Other: NORMAL CONDITION
- UNDERSTATED CONDITION: It involves an illusion with virtual reality where the patients perform a lumbar extension until the onset of pain and the feel a 10% less movement in the VR (understated visual feedback)
  Interventions: Other: UNDERSTATED CONDITION
- OVERSTATED CONDITION: It involves an illusion with virtual reality where the patients perform a lumbar extension until the onset of pain and the feel a 10% more movement in the VR (understated visual feedback)
  Interventions: Other: OVERSTATED CONDITION

INTERVENTIONS:
Other: NORMAL CONDITION — They perform 3 lumbar extensions until the onset of pain without virtual reality
  Groups: NORMAL CONDITION
Other: UNDERSTATED CONDITION — They perform 3 lumbar extensions until the onset of pain using the virtual reality. In this condition, they feel that they are moving a 10%less than they are really moving.
  Groups: UNDERSTATED CONDITION
Other: OVERSTATED CONDITION — They perform 3 lumbar extensions until the onset of pain using the virtual reality. In this condition, they feel that they are moving a 10% more than they are really moving.
  Groups: OVERSTATED CONDITION

SUMMARY:
This study investigates the potential to modify movement-evoked pain in individuals with chronic low back pain (LBP) by manipulating visual proprioceptive feedback through virtual reality (VR). Fifty patients with non-specific chronic LBP are planned to participate. Participants perform lumbar spine extension until pain onset under three conditions: accurate visual feedback (control), feedback showing 10% less movement (E-), and feedback showing 10% more movement (E+). Lumbar range of motion (ROM) is measured using a 3-space Fastrack motion analysis system. The study also explores whether individuals with higher pain levels, kinesiophobia, disability, or catastrophising are more susceptible to VR feedback manipulation. Pain thresholds, pain intensity, kinesiophobia, disability, and catastrophising levels are assessed.

DETAILED DESCRIPTION:
This study explores the potential to influence movement-evoked pain in individuals with chronic low back pain (LBP) by altering visual proprioceptive feedback using virtual reality (VR). The researchers aim to understand whether manipulating visual feedback can change pain perception and movement behavior. A total of 50 patients with non-specific chronic LBP are expected to participate.

Participants will perform lumbar spine extension movements until the point of pain onset under three experimental conditions: (1) without virtual reality (control); (2) underestimated movement feedback (E-), where the VR shows 10% less movement than performed; and (3) overestimated movement feedback (E+), where the VR depicts 10% more movement than performed. These manipulations aim to investigate how changes in perceived movement affect pain perception and range of motion.

The lumbar range of motion (ROM) is objectively measured using a 3-space Fastrack motion analysis system to ensure precise tracking of physical movements. Additionally, the study examines whether psychological factors, such as pain intensity, kinesiophobia (fear of movement), disability, and catastrophising (exaggerated negative mental set about pain), influence susceptibility to VR feedback manipulation.

To provide a comprehensive assessment, participants' pain thresholds, pain intensity levels, kinesiophobia, disability, and catastrophising tendencies are measured through validated tools. By combining physical and psychological evaluations, the study aims to identify potential subgroups of patients who might benefit most from VR-based interventions and shed light on the mechanisms through which visual feedback alters pain perception and movement behavior in chronic LB

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes.
* Aged between 18 and 65 years.
* Diagnosed with non-specific chronic low back pain (according to the European COST B13 guidelines).
* Presence of lumbar extension limitation.

Exclusion Criteria:

* Diagnosis of a spinal tumor.
* Presence of a spinal infection or fracture.
* Diagnosed systemic diseases.
* Diagnosis of fibromyalgia.
* Presence of cauda equina syndrome.
* History of prior spinal surgery.
* Musculoskeletal injuries of the lower extremities (including: sciatica; radiating pain in the lower extremities; symptoms of numbness or weakness in the lower extremities)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic low back pain
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
MOVEMENT EVOKED PAIN THRESHOLD | Baseline (pre-intervention) and immediately post-intervention (at 50 minutes).
  The maximum lumbar range of movement without pain was measured in each condition using a 3-Space Fastrack motion analysis system.
Pain Intensity | Baseline (pre-intervention) and immediately post-intervention (at 50 minutes).
  The pain intensity perceived by participants is measured using the Numeric Pain Rating Scale (NPRS-11)

SECONDARY OUTCOMES:
Fear of movement | Baseline (pre-intervention) and immediately post-intervention (at 50 minutes).
  The investigators will use the reliable and validated Spanish version of the Tampa Scale for Kinesiophobia (TSK), which consists of 11 independent phrases rated on a 4-point scale (1 = totally disagree to 4 = totally agree). Higher scores indicate higher levels of fear of movement.
Catastrophizing | Baseline (pre-intervention) and immediately post-intervention (at 50 minutes).
  The validated Spanish version of the Pain Catastrophizing Scale (PCS) will be applied, which has demonstrated internal consistency, test-retest reliability, and sensitivity to change. The PCS comprises 13 items rated on a 5-point scale from 0 (never) to 4 (always) that measure 3 components of catastrophising: rumination, magnification, and helplessness. Higher scores indicate greater pain-related catastrophising.
Disability | Baseline (pre-intervention) and immediately post-intervention (at 50 minutes).
  The degree of disability is measured using the validated and reliable Spanish version of the Roland-Morris Questionnaire (RMQ), which consists of 24 items whose scores range from 0 (no disability) to 24 (maximum disability)

CONTACTS AND LOCATIONS:
Locations (1):
- Arnau de Vilanova Hospital, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Harvie DS, Broecker M, Smith RT, Meulders A, Madden VJ, Moseley GL. Bogus visual feedback alters onset of movement-evoked pain in people with neck pain. Psychol Sci. 2015 Apr;26(4):385-92. doi: 10.1177/0956797614563339. Epub 2015 Feb 17. PMID 25691362